CLINICAL TRIAL: NCT03084016
Title: Exhaled Breath Biomarkers in Acute Asthma: A Feasibility Study
Brief Title: Asthma Breath Biomarker Assessment
Acronym: ABBA
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 197935
Record Dates: First submitted 2017-03-06; First posted 2017-03-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Asthma Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute asthma exacerbation: Recruited in secondary care when presenting with acute asthma exacerbation.
- At risk of acute asthma exacerbation: Recruited in outpatient clinics. Acute exacerbation within the previous 12 months.

SUMMARY:
This study aims to assess the feasibility of capturing data on exhaled breath compounds during an acute asthma exacerbation. In addition to assessing the feasibility of such a study the investigators will collect data on exploratory outcomes including the ability of breath biomarkers to distinguish between controlled and exacerbated states and their ability to differentiate between triggers of exacerbation.

DETAILED DESCRIPTION:
This will be a longitudinal observational study in which the investigators assess the ability to capture information on volatile organic compounds in exhaled breath during an acute asthma exacerbation using two different approaches:

A) Recruitment and assessment of patients in secondary care during an acute exacerbation of their asthma; patients to be re-assessed once their asthma is stable and controlled.

B) Recruitment of clinically stable outpatients who are at increased risk of exacerbation by virtue of having had an acute exacerbation within the previous 12 months. Participants to be followed for a period of up to 12 months; assessed in the event of an exacerbation; and re-assessed once controlled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Aged 18 or above
3. Able to provide informed consent
4. A confirmed asthma diagnosis requiring treatment with inhaled bronchodilator therapy +/- inhaled corticosteroids.
5. Non-smoker (or ex-smoker of 6 months or more with a less than 10 pack year history).
6. Current exacerbation or exacerbation within the previous 12 months.
7. Within 24 hours of having presented to acute secondary care (applicable to current exacerbation only)

Exclusion Criteria:

1. Major chronic cardiorespiratory disease other than asthma
2. Significant comorbid condition
3. Receiving maintenance oral corticosteroid therapy or other immunosuppressant or immunomodulatory therapy (including biologics)
4. Pregnant
5. Participating in a clinical trial of an investigational medicinal product (CTIMP).
6. Unable to speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18+ with asthma diagnosis meeting British Thoracic Society guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Study feasibility - recruitment | 18 months
  Recruitment rate
Study feasibility - assessment | 18 months
  Percentage of participants who experience an exacerbation, contact the study team and complete an assessment
Study feasibility - patient acceptability | 18 months
  Patient acceptability of breath capture devices (assessed by questionnaire)

SECONDARY OUTCOMES:
Breath profile of exhaled volatile organic compounds (VOCs). | 12 months
  A profile of VOCs in exhaled breath obtained through gas chromatography-mass spectrometry during asthma exacerbation and when stable.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wilson, Study Director — University of East Anglia
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PhD thesis — https://ueaeprints.uea.ac.uk/id/eprint/80211/